CLINICAL TRIAL: NCT00278434
Title: An Exploratory Clinical Trial of Zoledronic Acid in Women With CIN 2/3 or 3
Brief Title: Zoledronate in Treating Patients With Cervical Intraepithelial Neoplasia 2/3 or 3
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Accrual was insufficient to meet study endpoints
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDR0000460044; UCSF-03421; UCSF-H7810-25693-01; UCSF-H7810-25693-02A
Record Dates: First submitted 2006-01-16; First posted 2006-01-18 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Cervical Cancer; Precancerous Condition
Keywords: cervical cancer; cervical intraepithelial neoplasia grade 2; cervical intraepithelial neoplasia grade 3
MeSH Terms: conditions — Uterine Cervical Neoplasms; Precancerous Conditions; Uterine Cervical Dysplasia | interventions — Zoledronic Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Zoledronate (Experimental): 100 cc of saline with 4 mg of zoledronate intravenous (IV), over 20 minutes, for 3 doses one week apart
  Treatment repeats every 21 days (one course) for up to 3 courses. In week 8, patients undergo surgical resection comprising loop excision or cone biopsy.
  After completion of study treatment, patients are followed at week 10 by telephone.
  Interventions: Drug: Zoledronate
- Saline (Placebo Comparator): 100 cc of saline IV, over 20 minutes, for 3 doses one week apart
  Treatment repeats every 21 days (one course) for up to 3 courses. In week 8, patients undergo surgical resection comprising loop excision or cone biopsy.
  After completion of study treatment, patients are followed at week 10 by telephone.
  Interventions: Other: Placebo (Saline)

INTERVENTIONS:
Drug: Zoledronate
  Arms: Zoledronate
Other: Placebo (Saline)
  Arms: Saline

SUMMARY:
RATIONALE: Chemoprevention is the use of certain drugs to keep tumors from forming, growing, or coming back. Zoledronate may prevent the growth of cervical cancer by blocking blood flow to cervical intraepithelial neoplasia cells. The use of zoledronate may keep cancer from forming.

PURPOSE: This randomized is studying how well zoledronate works in treating patients with cervical intraepithelial neoplasia 2/3 or 3.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess clinical response, in terms of lesion size and histological grade, of oledronate in patients with cervical intraepithelial neoplasia 2/3 or 3.

OUTLINE: This is a randomized, placebo-controlled, double-blind, pilot study. Patients are stratified according to degree of cervical intraepithelial neoplasia (CIN) (CIN2/3 vs CIN3). Patients are randomized to 1 of 2 treatment arms.

* Zoledronate: 100 cc of saline with 4 mg of Zoledronate intravenous (IV), over 20 minutes, for 3 doses one week apart
* Placebo: 100 cc of saline (IV), over 20 minutes, for 3 doses one week apart

In both arms, treatment repeats every 21 days for up to 3 courses. In week 8, patients undergo surgical resection comprising loop excision or cone biopsy.

After completion of study treatment, patients are followed at week 10 by telephone.

PROJECTED ACCRUAL: A total of 44 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Biopsy confirmed cervical intraepithelial neoplasia (CIN) 2/3 or 3

  * Planning loop excision or cone biopsy
  * Diagnosis within 2 months prior to study entry
  * Standard histological grading according to Richart
* Visible lesion by colposcopy

  * No unsatisfactory colposcopy or lesions extending into the endocervical canal that cannot be visualized entirely by colposcopy
* No suspicion of invasive cervical cancer by cytology, histology or colposcopy
* No cytologic evidence of glandular atypia or dysplasia

PATIENT CHARACTERISTICS:

* Creatinine normal
* Screening laboratory values within normal range (e.g., complete blood count, liver function tests, renal panel, and electrolytes)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to read and speak English or Spanish
* No known hypersensitivity to bisphosphonates
* Not immunocompromised
* No known HIV positivity
* No aspirin-sensitive asthma due to association of bisphosphonates with bronchoconstriction
* No unexplained abnormal vaginal bleeding

PRIOR CONCURRENT THERAPY:

* No concurrent loop diuretics, aminoglycosides, other nephrotoxic drugs, immunosuppressive drugs, or other investigational agents

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2005-04; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Impact of Zoledronic Acid (ZA) on clinical response | 10 weeks from start of treatment
  The primary objective is to determine whether Zoledronic Acid (ZA), when given to women with CIN 2/3 or 3 for two months prior to surgical excision, has a measurable impact on clinical response (lesion size and histological grade).

CONTACTS AND LOCATIONS:
Overall Officials: Karen Smith-McCune, MD, PhD, Study Chair — University of California, San Francisco
Locations (1):
- UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California, United States